CLINICAL TRIAL: NCT07406126
Title: Y90 Radioembolization as Neoadjuvant Therapy for Potentially Resectable Patients With Colorectal Liver Metastases: Immune Markers Evaluation, Impact on Circulating Tumor DNA and Personalized Dosimetry Approach
Brief Title: Yttrium-90 Radioembolization Neoadjuvant Therapy With Immune Marker Profiling and Dosimetry for Potentially Resectable Patients With Colorectal Liver Metastases
Acronym: YRENE
Status: Not yet recruiting | Type: Observational
Sponsor: Fernando Gómez Muñoz (Other)
Collaborators: Instituto de Investigacion Sanitaria La Fe (Other); Boston Scientific International S.A. (Unknown)
Responsible Party: Sponsor-Investigator, Fernando Gómez Muñoz, Principal Investigator, MD, PhD, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Other Study IDs: GIBI2^30- YRENE
Record Dates: First submitted 2025-12-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Liver Metastases (CRCLM); Unresectable Colorectal Liver Metastases
Keywords: Unresectable Colorectal Liver Metastases; Potentially resectable patient; neoadjuvant therapy; Immune Marker Profiling; circulating tumor DNA; personalized dosimetry approach; Insufficient future liver remnant; Observational; multicenter; prospective; YRENE; TARE; TheraSphere®; Yttrium-90; Transarterial Radioembolization; primary colon adenocarcinoma; primary rectum adenocarcinoma; Unfavourable tumor location; metastatic disease; FOLFOX 6
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Yttrium-90 Radioembolization with standard systemic therapy — Yttrium-90 microspheres are administered through the hepatic artery which supplies blood to tumor tissue (the portal vein supplies blood to the normal hepatic tissue). The microspheres are trapped in the vasculature of the tumor due to arteriolar capillary blockage where they exert a local radiotherapeutic effect. In clinical use, the glass microspheres remain permanently trapped in the vasculature where the isotope decays to infinity leaving background radiation with no therapeutic value. This procedure is combined with standard systemic therapy per routine clinical practice.

SUMMARY:
This is a observational, prospective, single arm, proof of concept study to assess safety, feasibility, and potential efficacy of combining Yttrium-90 transarterial radioembolization(TARE) with standard systemic therapy in clinical practice for potentially resectable patients with colorectal liver metastases (CRLM). Alternatively, resectability will also be evaluated. The investigators hypothesize that by applying this approach, higher local control and resection rates can be achieved (typically below 13% for patients who are initially deemed unresectable). Additionally, this treatment option is expected to help delay or reduce the need for (a switch in) systemic treatment and eventually improve survival in patients with liver metastases that are not resectable. All studies reporting the results of TARE at ablative doses are retrospective cohort studies or cases series. Prospective data is needed to expand the indications and reimbursement of radioembolization.

Other objectives of the study are:

* To calculate the resection rate in patients undergoing the combined approach.
* To evaluate immune markers in peripheral blood and resected metastases.
* To formulate the first concept of an algorithm, enable to deliver personalized AI assisted dosimetry.
* To assess potential role of circulating tumor DNA (ctDNA) in evaluation of patient prognosis and follow up.
* To determine the grade of necrosis at the time of resection and correlate with the absorbed dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary adenocarcinoma of the colon or rectum
* Potentially resectable colorectal liver metastases, with limiting factors for resection including:

  1. Insufficient future liver remnant.
  2. Unfavorable tumor location (e.g. involvement of a major vessel and/or bile duct)/ large size and/ or number of lesions, which limit resection with R0 margins and requires downsizing of the metastases
* No or limited extrahepatic metastatic disease (limited extrahepatic disease should be amenable to eradicate with locoregional therapies as per multidisciplinary discussion of surgeons, radiation oncologists and interventional radiologists)
* Patient should match standard 90Y radioembolization inclusion criteria:

  1. Signed informed consent;
  2. Age ≥ 18 years;
  3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
  4. Life expectancy of ≥ 3 months;
  5. Measurable target tumors in the liver according to RECIST 1.1
* Laboratory parameters: eGFR >45/mL/min/1.73 m2; albumin > 3.0 g/dl, normal bilirubin (unless Gilbert syndrome); aminotransferase (ALAT/ASAT) <3.0 ULN

Exclusion Criteria:

* Life expectancy ≤3 months
* Patient initially eligible for surgery or thermal ablation of the liver metastases
* Progressive extra-hepatic disease
* Active extra-hepatic disease that cannot be treated
* Life-threatening extra-hepatic disease (i.e. dialysis, unresolved diarrhea, serious unresolved infections (HIV, HBV, HCV etc.))
* Uncorrectable coagulopathy
* Contraindication for angiography or MRI
* Significant toxicities due to prior cancer therapy that have not resolved before the initiation of the study; if the investigator determines that the continuing complication will compromise the safe treatment of the patient
* Any surgical contraindication
* Ascites
* Expected difficulties for safe execution of TARE based on pretreatment Tc99m-MAA imaging, including;
* Flow to extra-hepatic vessels not correctable by reposition of catheter or embolization Uncorrectable estimated dose to the lungs >30Gy in a single administration or >50Gy cumulatively
* Uncorrectable estimated dose to the untreated liver of >70Gy
* Estimated average dose to the viable tumor volume <200Gy
* Prior liver radiotherapy
* Severe portal hypertension
* Second primary malignancy within the past 5 years, other that adequately treated non-melanoma skin cancer, carcinoma in situ of any organ or second primary colorectal cancer
* Unresectable primary tumor in situ;
* Other serious comorbidity or any other condition, that renders patients unsuitable for the study treatment
* Pregnancy, lactation or refusal to use adequate contraceptive measures
* History of allergic reaction to any components of the treatment that cannot be medically corrected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (N = 30) with insufficient FLR and patients with unfavorable lesion location, size and/ or number, requiring downsizing of metastases in order to achieve R0 resection will be discussed at the respective local multidisciplinary teams (MDT) meetings. Patients can be included if they are found suitable for TARE and surgery based on a liver MRI, contrast enhanced CT or PET-CT and clinical and laboratory results. Patients are allowed to undergo other local liver treatments (e.g. ablation) in combination with TARE, as long as all liver metastasis are locally treated to achieve R0 resection. Patients are not allowed to use systemic chemotherapy two weeks prior and two weeks post TARE. Target therapies have to be stopped at least 4 weeks prior to TARE.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Monitoring for adverse events related to the procedure. | From 90Y radioembolization (week 2-4) to the end of study at 30 weeks
  Evaluate the safety of combining neoadjuvant ablative dose 90Y radioembolization with standard systemic therapy in patients with CRLM. Safety assessments will include monitoring for adverse events related to the procedure.
Evaluate the safety related to the procedure by measuring changes in Liver function values in blood. | From 90Y radioembolization (week 2-4) to the end of study at 30 weeks
  To evaluate hepatic safety after neoadjuvant ablative-dose Yttrium-90 radioembolization combined with standard systemic therapy in patients with CRLM changes in laboratory biomarkers will be compared with baseline values and subsequent assessments.
  Biomarkers and Units of Measure:
  - Liver Function Markers: Bilirubin (mg/dL), Albumin (g/dL), Aspartate Aminotransferase (AST) (U/L), Alanine Aminotransferase (ALT) (U/L), Gamma-Glutamyl Transferase (GGT) (U/L), Alkaline Phosphatase (FA) (U/L), Cholinesterase (ChE) (U/L), Lactate Dehydrogenase (LDH) (U/L)
Evaluate the safety related to the procedure by measuring changes in Liver function values in blood. | From 90Y radioembolization (week 2-4) to the end of study at 30 weeks
  To evaluate hepatic safety after neoadjuvant ablative-dose Yttrium-90 radioembolization combined with standard systemic therapy in patients with CRLM changes in laboratory biomarkers will be compared with baseline values and subsequent assessments.
  Biomarkers and Units of Measure:
  Inflammatory Marker: C-reactive protein (CRP) (mg/L) Renal Function Marker: Creatinine (mg/dL)
Evaluate the safety related to the procedure by measuring changes in Liver function values in blood. | From 90Y radioembolization (week 2-4) to the end of study at 30 weeks
  To evaluate hepatic safety after neoadjuvant ablative-dose Yttrium-90 radioembolization combined with standard systemic therapy in patients with CRLM changes in laboratory biomarkers will be compared with baseline values and subsequent assessments.
  Biomarkers and Units of Measure:
  Composite Liver Function Scores: Albumin-Bilirubin (ALBI) score (unitless), Albumin-Bilirubin (ALBI) grade (ordinal scale)
Evaluate the safety related to the procedure by measuring changes in tumor markers in blood. | From 90Y radioembolization (week 2-4) to the end of study at 30 weeks
  Evaluate the safety of combining neoadjuvant ablative dose 90Y radioembolization with standard systemic therapy in patients with CRLM by assessing tumor markers in blood: Carcinoembryonic antigen (CEA) and CA 19-9.
Evaluate the quality of Life After Liver Resection Assessed by FACT-C (Version 4) Following 90Y Radioembolization | From 90Y radioembolization (week 2-4) to the end of study at 30 weeks
  Evaluate the safety of combining neoadjuvant ablative dose 90Y radioembolization with standard systemic therapy in patients with CRLM. Safety assessments will include assessing overall well-being of the patients focus on quality of life after liver resection.
  Outcome Measure: Change in Functional Assessment of Cancer Therapy-Colorectal (FACT-C, Version 4) total score from baseline to 30 weeks. The FACT-C (Version 4) total score and each subscale will be analyzed as independent measures to evaluate longitudinal changes in overall well-being and postoperative recovery after liver resection, characterizing treatment-related safety and tolerability.
  Quality-of-Life Instrument:
  Functional Assessment of Cancer Therapy-Colorectal (FACT-C, Version 4): Total score and subscale scores (Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Colorectal Cancer Subscale), reported according to standard scoring guidelines.
Evaluate the efficacy of the procedure by tumor response rate assessed by means of RECIST 1.1 | From week 0 to resection, progression or week 26-28
  Efficacy assessments will include tumor response rate assessed by means of RECIST 1.1. Baseline efficacy imaging scans will be conducted during the screening phase. Efficacy assessment scans will follow standard-of-care clinical management guidelines, occurring every 8 weeks (with a variance of +/- 1 week) post-inclusion until resection or until progression.
Evaluate the efficacy of the procedure: pathologic response assessment on the resected specimens. | From week 0 to resection, progression or week 26-28
  Efficacy assessments will include tumor response rate assessed by means of RECIST 1.1. It will be of capital interest the pathologic response assessment on the resected specimens.

SECONDARY OUTCOMES:
Resection rate in patients undergoing the combined approach | week 18-20 and week 26-28
  It will indicate the percentage of patients who ultimately proceed to surgical resection of their liver metastases after receiving TARE as part of the neoadjuvant therapy. The decision of resection will be taken in the respective multidisciplinary meetings of each participating center.
Cellular population quantification on peripheral blood samples: leukocytes, neutrophils, lymphocytes, monocytes, eosinophils and basophils. | Week 0, 6, 8 and 16
  Microbial fuel cell procedure will be performed on peripheral blood samples within the first 24-36 hours after collection. Bulk lysis technique will be done with the aim to concentrate leukocytes and, later, to detect minority populations. The quantification of each population will be performed in percentage and in absolute count, estimating the cells per microliter from the leukocyte value obtained in the complete blood count (CBC). In fact, a CBC will be done obtaining the percentages and absolutes values of neutrophils, lymphocytes, monocytes, eosinophils and basophils. Neutrophil-to-lymphocyte and lymphocyte-to-monocyte ratios will be estimated.
Inflammatory interleukines IL-6, IL-10 and IFN-γ quantification: | Week 0, 6, 8 and 16
  Cytokines IL6 and IL10 levels
Intratumoral T Cells Infiltration in biopsies and resected tumors. | week 0, week 18/20 and week 26/28
  The density of each tumor-infiltrating immune cell (CD3 and CD8) will be assessed in biopsies and resected tumors.
PERSONALIZED AI ASSISTED DOSIMETRY evaluation | week 0 to 26-28
  AI assisted dosimetry will be evaluated by the creation of a predictive model to assess treatment outcome based on planned and post-treatment high precision dose estimates. A prediction model based on corrected planning SPECT/CT and post-treatment PET/CT.
ctDNA analysis: Identification of genetic alterations and circulating tumor DNA (ctDNA) monitoring through digital droplet PCR | week 6, 8, 12, 16, 22 and 30
  Sample collection and Nucleic acid isolation will be performed by means of Formalin-fixed paraffin embedded (FFPE) tumor biopsies (metastases). Two 10 mL Cell-Free DNA BCT ® CE (Streck) tubes of peripheral blood will be extracted for liquid biopsy studies. In FFPE tumour by NGS colorectal cancer cells are characterized by the acquisition of molecular alterations responsible for tumor development and progression. Digital droplet PCR (ddPCR) has emerged as an ultra-sensitive approach with various applications in the molecular diagnosis of tumors especially in liquid biopsy studies. KRAS, NRAS and BRAF mutation detection will be carried out.
Macroscopic determination of the grade of necrosis | week 18/20 and week 26/28.
  the grade of necrosis will be analyzed through Histochemical staining of histological samples: standard hematoxylin-eosin staining. Staining of non-tumor liver with at least: Masson's trichrome and reticulin.
Determination of the grade of necrosis: Microscopic study. | week 18/20 and week 26/28.
  The Microscopic report will include the number of nodules, size, distance to margin in mm, tumor regression grade and the lesions observed in the non-tumor liver parenchyma in resected tumors. With the presence or absence of viable tumor cells, it is advisable to report on the presence or absence of: Fibrosis, Necrosis, specifying whether it is of the normal or infarct-type and mucous extracellular.
Evaluation of Post-treatment liver damage: Microscopic study | week 18/20 and week 26/28.
  Post-treatment liver damage: Presence and severity of steatosis, steatohepatitis and lesions related to the sinusoidal obstruction syndrome will be reported.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Provincial de Castellón, Castelló
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario y Politécnico la Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the published results will be shared with qualified researchers upon reasonable request. Data will be available after publication for a period of 5 years. Requests should be directed to GIBI230@iislafe.es. Access will be provided after approval of a proposal and execution of a data use agreement.
Time Frame: Data will be available after publication for a period of 5 years.
Access Criteria: Qualified researchers upon reasonable request directed to GIBI230@iislafe.es.

REFERENCES:
- [Background] Alsultan AA, et al. Dose-Response and Dose-Toxicity Relationships for Glass 90Y Radioembolization in Patients with Liver Metastases from Colorectal Cancer. J Nucl Med. 2021 Nov;62(11):1616-1623.
- [Background] Mulcahy MF. et al. EPOCH Investigators. Radioembolization With Chemotherapy for Colorectal Liver Metastases: A Randomized, Open-Label, International, Multicenter, Phase III Trial. J Clin Oncol. Dec 10;39(35):3897-3907 (2021).
- [Background] Torkian P. et al. Cancer Immunology: Impact of Radioembolization of Hepatocellular Carcinoma on Immune Response Modulation. AJR Am J Roentgenol. Jun;220(6):863-872 (2023)
- [Background] Garin E, et al. DOSISPHERE-01 Study Group. Personalised versus standard dosimetry approach of selective internal radiation therapy in patients with locally advanced hepatocellular carcinoma (DOSISPHERE-01): a randomised, multicentre, open-label phase 2 trial. Lancet Gastroenterol Hepatol. Jan;6(1):17-29 (2021).
- [Background] Simmonds, P. C. et al. Surgical resection of hepatic metastases from colorectal cancer: a systematic review of published studies. British journal of cancer 94, 982-999, doi:10.1038/sj.bjc.6603033 (2006).
- [Background] De Greef, K. et al. Multisciplinary management of patients with liver metastasis from colorectal cancer. World journal of gastroenterology 22, 7215-7225, doi:10.3748/wjg.v22.i32.7215 (2016)
- See also: American Cancer Society. Key Statistics for Colorectal Cancer. — https://www.cancer.org/cancer/colon-rectal-cancer/about/key-statistics.html